CLINICAL TRIAL: NCT02274584
Title: Safety and Efficacy Evaluation of 4th Generation Safety-engineered CAR T Cells Targeting Relapsed and Refractory CD30 Positive Lymphomas
Brief Title: CAR T Cells Targeting CD30 Positive Lymphomas (4SCAR30273)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Jun Zhu, Director, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30273-4SCAR
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Lymphomas
Keywords: Hodgkin's lymphoma; Anaplastic large cell lymphoma; CD30 positive lymphoma; Peripheral T/Natural Killer (NK) cell lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR T cells (Experimental): Autologous 4th generation anti-CD30 CAR T cells
  Interventions: Genetic: Anti-CD30 CAR T cells

INTERVENTIONS:
Genetic: Anti-CD30 CAR T cells — Autologous 4th generation withdrawal lentiviral-transduced anti-CD30 CAR T cells

SUMMARY:
Currently, a majority of lymphomas cannot be cured by standard chemo-radiotherapy. Cluster of differentiation antigen 30 (CD30) is expressed in many lymphoma subtypes, such as Hodgkin lymphoma (HL) and anaplastic large cell lymphoma (ALCL). CD30 represents a very attractive target for chimeric antigen receptor (CAR)-based immune cell therapy. This study will evaluate a novel 4th generation CD30 CAR engineered with a self-withdrawal mechanism (FKBP-iCasp9) for both efficacy and safety evaluation in lymphoma patients.

DETAILED DESCRIPTION:
A large number of lymphoma patients exhaust current treatment options and die from the disease. Innovative therapy is urgently needed. Chimeric antigen receptor (CAR)-modified T cells have demonstrated unprecedented successes in treating even late stage cluster of differentiation antigen 19 (CD19) positive B cell malignancies. Besides CD19 lymphomas, many lymphomas are CD30 positive and therefore, CD30-CAR T cells may prove to be effective in treating such patients. We have developed several generations of CD30 CARs. Preclinical studies have demonstrated effective killing of CD30 target cells. In this study, two versions of CD30 CARs, both of which are 4th generation CARs with a self-withdrawal mechanism (FKBP-iCasp9), will be evaluated in CD30 lymphoma patients. The primary goal is safety assessment including cytokine storm response and any other adverse effects. In addition, tumor targeting and disease status after treatment will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CD30(+) lymphoma patients proved by immuno-histochemistry (IHC) or Flow-cytometry.
* Not eligible for autologous stem-cell transplantation (ASCT) or relapsed after ASCT.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Age≥18.
* Pulse oximetry of > 90% on room air.
* Adequate hepatic function, defined as alanine transaminase (ALT) <3 x upper limit of normal (ULN), aspartate aminotransferase (AST) <3 x ULN; serum bilirubin and alkaline phosphatase <2 x ULN.
* Adequate renal function, defined as serum creatinine <2.0mg/dl.
* Adequate heart function with LVEF≥50%
* Hb≥80g/L
* Measurable disease can be identified.
* Life expectancy ≥3 months.
* Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 1 year after the study is concluded. The male partner should use a condom.
* Patients must sign an informed consent.

Exclusion Criteria:

* Uncontrolled active infection.
* Active infection with hepatitis B virus (HBV), hepatitis C virus (HCV).
* HIV positive
* Pregnant or lactating.
* Currently enrolled in another clinical trial.
* Concurrent use of systemic steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events. | 2 years.
  Determine the toxicity profile of the 4th generation CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Survival time of Anti-CD30 CAR T cells in vivo. | 2 years.
  Measure the survival of 4th generation CAR T cells transduced with the anti-CD30 lentiviral vector.
Response rates to the 4th generation CAR T cells. | 2 years.
  Describe the response rates of patients treated with 4th generation CAR T cells, including partial remission (PR), complete remission (CR), stable disease (SD) and progressive disease (PD).
Survival time of the patients. | 2 years.
  Evaluate the survival time of the patients treated with the 4th generation CAR T cells, including progression free survival (PFS) and overall survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- University of Florida, Gainesville, Florida, United States
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China